CLINICAL TRIAL: NCT04622566
Title: A Phase II Study of Neoadjuvant Lenvatinib and Pembrolizumab in Resectable Mucosal Melanoma
Brief Title: Lenvatinib and Pembrolizumab in Resectable Mucosal Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Director of Renal carcinoma and Melanoma Department in Bejing Cancer Hospital, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK59132
Record Dates: First submitted 2020-10-28; First posted 2020-11-10 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Mucosal Melanoma; Neoadjuvant Treatment
Keywords: pembrolizumab; Lenvatinib
MeSH Terms: interventions — lenvatinib; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Lenvatinib and Pembrolizumab in Resectable mucosal Melanoma. (Experimental)
  Interventions: Drug: Lenvatinib, Pembrolizumab

INTERVENTIONS:
Drug: Lenvatinib, Pembrolizumab — After enrollment, patients receive pembrolizumab 200 mg via IV infusion on Day 1 of each 3-week cycle for 6 weeks; Lenvatinib 20mg orally once daily for 6 weeks. Patients conduct surgery within 1-4 weeks after the last dose of Pembrolizumab and Lenvatinib. After complete surgery, Pembrolizumab will be as adjuvant treatment for up to 15 cycles, 200mg IV on day 1 of every 21 day-cycles.
  Other Names: Biological: Pembrolizumab IV infusion Other Names: MK-3475; KEYTRUDA®; Drug: Lenvatinib Oral capsule Other Names: MK-7902; E7080; LENVIMA®

SUMMARY:
This study is a randomized ,single center clinical study which is designed to investigate whether combination of Pembrolizumab with Lenvatinib could improve pCR rate and consequent survival in resectable mucosal melanoma.

All the eligible patients were assigned to receive Lenvatinib once a day (QD) for 6 weeks plus pembrolizumab on Day 1 of each 21-day cycle (Q3W) concurrently on days 1 and 22, followed by surgery and 18 cycles of Pembrolizumab 200mg q3w of adjuvant phase.

DETAILED DESCRIPTION:
Mucosal melanoma is a rare type of melanoma in Caucasian population and a dominate subtype in Asia, which generally carries a worse prognosis than cutaneous melanoma. Surgery remains the primary therapeutic intervention for mucosal melanoma, and neoadjuvant therapy is still needed which can lead to improvements in outcomes by surgical resectability, local control and organ preservation.

Immunotherapy has showed promising activity in advanced melanoma. However, PD-1 antibodies, both Pembrolizumab and Nivolumab, showed much poorer response to mucosal melanoma than to cutaneous melanoma.

Pembrolizumab showed modest objective response rate (ORR, 13%) in advanced mucosal melanoma in Chinese population (NCT02628067). Recent study also demonstrated that neoadjuvant therapy with one dose of Pembrolizumab could lead to pathological complete response (pCR) or major response in nearly 30% of resectable advanced melanoma and pCR was associated with reduced risk of recurrence and improved survival.

Lenvatinib is also a kinase inhibitor that inhibits the kinase activities of VEGFR1,2, 3 which has been approved by FDA for differentiated thyroid cancer, advanced renal cell carcinoma and hepatocellular carcinoma.

It is hypothesized that neoadjuvant Pembrolizumab in combination with Lenvatinib could result in higher anti-tumor activity with lower toxicity and prolong RFS and OS in high-risk resectable mucosal melanoma.

The study will assess the efficacy and safety of the combination Pembrolizumab and Lenvatinib as neoadjuvant treatment in resectable mucosal melanoma.

ELIGIBILITY:
Inclusion Criteria:

* 1. Be willing and able to provide written informed consent for the trial. 2. Be a male or female subject and is 18-75 years of age on day of signing informed consent.

  3. Have histologically or cytologically confirmed resectable mucosal melanoma. Only cases where a complete surgical resection with tumour-free margins can safely be achieved, as assessed by the surgeon, are defined as resectable.

  4. Newly diagnosed melanoma without any previous anti-cancer treatment 5. Patients must be able to provide a biopsy at baseline 6. Able to swallow and retain oral medication 7. Be medically fit enough to undergo surgery as determined by the treating medical and surgical oncology team 8. Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 10 days of treatment initiation.

  9. Demonstrate adequate organ function as defined in Table 1. All screening labs should be performed within 1 week prior to treatment initiation.

  10. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mmHg at screening and no change in antihypertensive medications within 1 week before treatment initiation.

  11. Males and female subjects of childbearing potential must be willing to use an adequate method of contraception, for the course of the study through 120 days after the last dose of study medication.

  12. (Female subject of childbearing potential) Have a negative urine or serum pregnancy test within 1 week prior to receiving the first dose of study medication. If the urine test is positive or borderline a serum pregnancy test will be required.

Exclusion Criteria:

* 1. Has a known additional malignancy that is progressing or requires active treatment, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.

  2. Has known central nervous system (CNS) metastases and/or carcinomatous meningitis.

  3. Has received any prior systemic anti-cancer treatment for melanoma 4. Has received prior lenvatinib 5. Has received prior therapy with an anti-PD-1 or anti-PD-L1 agent 6. Is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 4 weeks of the first dose of treatment in this current trial.

Note: subject should be excluded if he/she received an investigational agent with anti-cancer or anti-proliferative intent within the last 12 months.

7. Has received a live vaccine within 30 days of the first dose of study treatment.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., FluMist ®) are live attenuated vaccines, and are not allowed.

8. Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.

9. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 1 week prior to the first dose of trial treatment.

10. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).

11. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).

12. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis 13. Has an active infection requiring systemic therapy. 14. Has presence of gastrointestinal condition including malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.

15. Has had a major surgery within 4 weeks prior to initiation of treatment. Adequate wound healing after major surgery must be assessed clinically and have resolved completely.

16. Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula.

17. Has radiographic evidence of major blood vessel invasion/infiltration. The degree of tumor invasion/infiltration of major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.

18. Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study drug.

19. Has clinically significant cardiovascular disease within 12 months of the first dose of study intervention including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.

Note: Medically controlled arrhythmia would be permitted. 20. Has urine protein ≥1 g/24-hour. Note: Participants with >1+ proteinuria on urine dipstick will undergo 24-hour urine collection for quantitative assessment of proteinuria.

21. Has prolongation of QTc interval (calculated using Fridericia's formula) to >480 msec.

22. Has left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multi-gated acquisition scan (MUGA) or echocardiogram.

23. Has a history or current evidence of any condition, therapy, lab abnormality or other circumstance that might expose the subject to risk by participating in the trial, confound the results of the trial, or interfere with the subject's participation for the full duration of the trial.

24. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

25. Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of study medication.

26. Has a known hypersensitivity to the components of the study therapy or its analogs.

27. Has a known history of active TB (Bacillus Tuberculosis) Female participants who are breastfeeding are not eligible for enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2020-12-30 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate: defined as the percentage of subjects without alive tumor cells in the resected specimen post operation. | Approximately 10 weeks
  To evaluate pathological complete response (pCR) rate of Pembrolizumab combined with Lenvatinib as neoadjuvant therapy for resectable mucosal melanoma.

SECONDARY OUTCOMES:
1 year RFS (recurrence-free survival) rate per RECIST1.1 as Assessed by investigator | Approximately 1 year
  To evaluate1-year RFS rate of Pembrolizumab combined with Lenvatinib as neoadjuvant therapy for resectable mucosal melanoma.
Overall survival | Approximately 2 years
  OS is defined as the time from date of randomization to date of death from any cause. OS will be presented.
Incidence of AEs/SAEs | Approximately 2 years
  Adverse events (AEs) ; serious adverse events (SAEs); abnormal value of Lab test according to NCI-CTCAE V5.0

OTHER OUTCOMES:
The time from surgery completion to wound healing | Approximately 12 weeks
  To evaluate pembrolizumab with Lenvatinib as neoadjuvant treatment impact on surgery outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China